CLINICAL TRIAL: NCT06931990
Title: A Phase Ic/II Clinical Study to Explore the Safety, Tolerability, Efficacy, and Pharmacokinetics of Multiple Oral Doses of LT-002-158 Tablets in Chinese Adult Subjects With Atopic Dermatitis
Brief Title: A Study to Explore the Safety, Tolerability, Efficacy, and Pharmacokinetics of LT-002-158 Tablets in Chinese Adult Subjects With Atopic Dermatitis
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Leadingtac Pharmaceutical (Shaoxing) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LT2158CHN004
Record Dates: First submitted 2025-04-02; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Atopic Dermatitis (AD)
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LT-002-158 tablets low-dose group (Experimental)
  Interventions: Drug: LT-002-158 tablets
- LT-002-158 tablets high-dose group (Experimental)
  Interventions: Drug: LT-002-158 tablets

INTERVENTIONS:
Drug: LT-002-158 tablets — The subjects will orally administered LT-002-158 tablets once a day.

SUMMARY:
This study is an Ic/II phase clinical trial conducted in Chinese subjects with moderate to severe atopic dermatitis. The phase Ic study is a randomized, open label, parallel group design, mainly evaluating the safety and tolerability of LT-002-158 tablets in subjects with moderate to severe atopic dermatitis. The phase II study is a randomized, double-blind, placebo-controlled, parallel group design, with a single arm design for extended treatment, mainly exploring the efficacy of LT-002-158 tablets in the treatment of moderate to severe atopic dermatitis subjects.

ELIGIBILITY:
Inclusion Criteria:

1. When signing the informed consent form, the age range is 18 to 75 years old (including threshold), and there is no gender limit.
2. Body mass index (BMI) is between 17.5 and 40.0 kg/m2 (inclusive), with a weight of ≥ 45.0 kg.
3. Insufficient response or intolerance to topical corticosteroids (TCS) or topical calcineurin inhibitors (TCI) within the last 6 months of randomization; Insufficient response is defined as the failure to achieve and maintain remission or low disease activity (equivalent to vIGA 0=complete clearance to 2=mild) despite the use of a moderate to high efficacy TCS regimen (± TCI if applicable) for at least 28 days or the longest duration recommended in the drug prescription information (e.g. 14 days for super potent TCS), whichever is shorter.
4. Subjects must use topical moisturizers (moisturizers) daily for at least 7 consecutive days prior to the baseline visit. Participants should continue to use daily moisturizers during the study period.
5. Female and male participants with fertility and their partners had no fertility plans during the study period and within 6 months after the last dose, and agreed to take effective contraceptive measures.
6. Understand and voluntarily sign written informed consent; Willing and able to complete planned visits, treatments, examinations, and other procedures (such as dietary requirements, diary card recording, and collection) according to the requirements of the plan.

Exclusion Criteria:

1. Merge other skin diseases that may interfere with the study evaluation, such as psoriasis, tinea corporis, lupus erythematosus, etc.
2. Systemic anti infective therapy is required for active or chronic recurrent infections within the 4 weeks prior to the baseline visit.
3. Known or suspected to have a history of immune deficiency disease, other immune related diseases, invasive opportunistic infections or associated active tuberculosis.
4. History of severe or recurrent herpes virus infection, such as herpetic encephalitis, disseminated herpes, etc.
5. History of important organ transplantation (such as heart, lung, kidney, liver) or hematopoietic stem cell/bone marrow transplantation.
6. After inquiry, there is a history of lymphoproliferative diseases; Or currently suffering from malignant tumors or having a history of malignant tumors (excluding squamous cell carcinoma in situ of the skin, basal cell carcinoma, and cervical cancer in situ, which have achieved complete remission after radical treatment for more than 5 years without any signs of recurrence).
7. A family history of sudden death or long QT syndrome, or subjects with a history of congenital or drug-induced long QT syndrome.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment emergent Adverse Events | up to 42 days

SECONDARY OUTCOMES:
Area under the curve plasma concentration from time zero to last measurable concentration [AUC(0-last)] | up to 42 days
Maximum observed plasma concentration at steady state (Cmax,ss) | up to 42 days
Minimum observed plasma concentration at stead state (Cmin,ss) | up to 42 days